CLINICAL TRIAL: NCT06149039
Title: Study on Lymphocyte Subsets of Peripheral Blood in Patients With Nonmyopathic Dermatomyositis Complicated With Pulmonary Interstitial Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yanfeng Hou (Other)
Responsible Party: Sponsor-Investigator, Yanfeng Hou, professor, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Other Study IDs: YXH2022ZX03223
Record Dates: First submitted 2023-11-13; First posted 2023-11-28 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Dermatomyositis
MeSH Terms: conditions — Dermatomyositis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Nonmyopathic dermatomyositis with interstitial lung disease
- Classical dermatomyositis with interstitial lung disease
- Rheumatic disease with interstitial lung disease in non-inflammatory myopathy
- Healthy adult

SUMMARY:
To detect the changes of lymphocyte subsets in peripheral blood of non-myopathic dermatomyositis with pulmonary interstitial disease, classical dermatomyositis with pulmonary interstitial disease, rheumatism with non-inflammatory myopathy with pulmonary interstitial disease and healthy adults among the 4 groups, and to detect the related cytokines secreted by lymphocyte subsets Th1,Th2 and Th17. Clinical features, distribution of peripheral lymphocyte subsets ratio and related cytokine content secreted by each lymphocyte subset were analyzed in each group, so as to explore the pathogenesis characteristics of nonmyopathic dermatomyositis complicated with pulmonary interstitial disease, in order to facilitate clinical guidance for diagnosis and treatment.

ELIGIBILITY:
Inclusion Criteria:

1. The experimental group met the diagnostic criteria of Sontheimer and was diagnosed as CADM with pulmonary interstitial disease.
2. Control group 1: The diagnosis was consistent with the diagnostic criteria of Bohan and Perter classification system, and it was confirmed that dermatomyositis was combined with pulmonary interstitial disease;
3. Control group 2: The diagnosis meets the classification criteria of systemic lupus erythematosus revised by the American College of Rheumatology (ACR) in 1997 and is confirmed as systemic lupus erythematosus combined with pulmonary interstitial disease, or the diagnosis meets the diagnostic criteria of rheumatoid arthritis introduced by ACR in 1987 or ACR in 2010 and is confirmed as rheumatoid arthritis combined with pulmonary interstitial disease.
4. Age 18-70 years old;
5. Have a good understanding of their own illness and physical condition, have self-knowledge, can communicate well with others;
6. Voluntarily join the study, understand the significance of the experiment and the indicators to be measured, and sign the informed consent.

Exclusion Criteria:

1. Severe infection: fever, cough, phlegm, sore throat, abdominal pain, diarrhea, carbuncle and other skin and soft tissue infection and other clinical manifestations, blood routine white blood cell count beyond the normal range (10×109/L);
2. Severe cardiovascular disease: including chronic heart dysfunction grade 3 or above and various arrhythmias;
3. Infectious diseases: hepatitis active stage, AIDS, syphilis, etc.
4. Tumor markers of patients suggest the possibility of tumor.
5. Patients with neuromuscular disease, inflammatory bowel disease, functional gastrointestinal disease;
6. The patient has other connective tissue diseases or disorders.

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients and healthy adults who meet inclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
T helper 1 cell | 2023-04-01 - 2024-06-30
  Th1 cells are a type of lymphocytes that can produce pro-inflammatory cytokines to support the body's immune response.
T helper 2 cell | 2023-04-01 - 2024-06-30
  Th2 is a T cell subset that can secrete Th2 type cytokines (such as interleukin IL-4, IL-5, IL-10 and IL-13, etc.), belonging to CD4+T cells.
T helper 17 cell | 2023-04-01 - 2024-06-30
  Th17 cells are an important subset of CD4+T lymphocytes, which can express specific transcription factor RORγT and secrete cytokine IL-17.

CONTACTS AND LOCATIONS:
Locations (1):
- Yanfeng Hou, Jinan, Shandong, China